CLINICAL TRIAL: NCT04439721
Title: Safety and Effectiveness of Donor γδT Cell Infusion to Prevent Relapsed/Refractory Leukemia Rescue Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: γδT Cell Infusion to Prevent Relapsed/Refractory Leukemia Rescue Relapse
Acronym: γδT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PG-γδT-001
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Leukemia, B-cell
Keywords: γδT; leukemia
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- γδT (Experimental): γδT,Infusion,iv,0.5×10^6-8×10^7γδT /kg,once.
  Interventions: Drug: γδT Cell infusion agent

INTERVENTIONS:
Drug: γδT Cell infusion agent — γδT

SUMMARY:
Safety and Effectiveness of Donor γδT Cell Infusion to Prevent Relapsed/Refractory Leukemia Rescue Relapse After Allogeneic Hematopoietic Stem Cell Transplantation

DETAILED DESCRIPTION:
γδT cells belong to the innate immune system and have a powerful anti-tumor effect. Leukemia patients transplanted with allogeneic hematopoietic stem cells have an important role in controlling leukemia recurrence. Although adoptive immunotherapy using in vitro expanded γδT cells has achieved significant results in patients with solid tumors, infusion of donor γδT cells in leukemia patients undergoing allogeneic hematopoietic stem cell transplantation to prevent leukemia recurrence has not been reported. . This clinical study intends to initially observe the safety and effectiveness of donor γδT cell infusion to prevent recurrence/refractory leukemia salvage allogeneic hematopoietic stem cell transplantation to further improve the transplantation effect of these patients

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia patients undergoing salvage allogeneic hematopoietic stem cell transplantation
* Age 10-65,Any gender
* Expected lifetime>3months
* ECOG 0-2
* DSA Negative
* Successful granulocyte implantation
* Liver and kidney function, heart and lung function meet the following requirements:①Creatinine≤1.5 ULN；②ALT/AST ≤5 ULN； ③Baseline oxygen saturation≥92%； ④Left ventricular ejection fraction≥50%
* Female subjects with fertility who had a negative pregnancy test within 48 hours before the infusion and were not breastfeeding; all subjects with fertility potential before enrolling in the study and throughout the study period until the last infusion Within 3 months, take adequate contraceptive measures
* Signing informed consent patients must be able to understand and be willing to participate in this study, and sign informed consent at the same time

Exclusion Criteria:

* Donor HBsAg or HBcAb positive and HBV DNA titer test is not within the normal reference value; donor or patient HCV antibody positive and peripheral blood HCV RNA positive; donor or patient HIV antibody positive; donor syphilis test positive
* Active central nervous system disease
* BMI index>35
* Allergic to DMSO
* Graft-versus-host disease
* Septic shock
* Systemic steroid therapy is required during cell infusion or cell collection, or there are conditions that researchers believe may require steroid therapy during blood collection or during infusion. In addition to cell collection or infusion, steroids for disease treatment are allowed, and inhaled steroids or hydrocortisone are also allowed for physiological replacement therapy in patients with adrenal insufficiency
* Participated in another clinical trial within 4 weeks before enrolling in the study, or intend to participate in another clinical trial throughout the study
* According to the judgment of the investigator, it does not meet the situation of cell preparation
* Circumstances considered by other researchers to be inappropriate

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the dose limiting toxicity (DLT) | 4 weeks after γδT infusion
  Toxicity will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale, version 5 and the number of patients experiencing DLT will be evaluated.
The incidence of serious adverse events (SAEs) | 4 weeks after γδT infusion
  The incidence of serious adverse events (SAEs) after γδT infusion

SECONDARY OUTCOMES:
Disease-free survival time(DFS) | about 2 years after γδT infusion
  γδT cell infusion treatment of CR/CRi patients from the beginning of γδT cell infusion treatment to the first disease recurrence or death from any cause
Overall survival (OS) | about 2 years after γδT infusion
  The time from the subject receiving γδT cell infusion treatment to death (for any reason)
Duration of remission after administration (DOR) | about 2 years after γδT infusion
  γδT cell infusion treatment has not reached CR/CRi before the treatment, the time from the first assessment of CR/CRi after administration to the first assessment of disease recurrence or progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Ph.D, Principal Investigator — Hematology，The First Affiliaated Hospital Of Soochow University
Locations (1):
- No.188 Shizi Street, Suzhou, Jiangsu, China